CLINICAL TRIAL: NCT05485493
Title: The Effectiveness of Internet-Based Solution Focused Short-Term Group Counseling on Emotional Eating Levels of Nursing Students
Brief Title: The Effect of Solution-focused Approach on Emotional Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Merve Saritas, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MSaritas
Record Dates: First submitted 2022-08-02; First posted 2022-08-03 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-08

CONDITIONS: Emotional Eating
Keywords: emotional eating; solution focused counseling; nursing student; body mass index
MeSH Terms: conditions — Emotional Eating

STUDY DESIGN:
Intervention Model Description: The research is a randomized controlled experimental model with a pretest posttest control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The counseling program is 6 sessions, and it is the sessions will last 60-90 minutes on average once a week and be conducted via online video-conference applications. The first session is informing group members about emotional eating and solution-oriented approach, determining members' goals and expectations. Second session; It aims to ensure that emotions are noticed, to clarify the goals with the miracle question technique, and to focus on the solution by getting away from the problems. In the third session; Exception questions focus on recognizing exceptional situations, strengths, and skills. In the fourth session; It is aimed to discuss the existing coping methods of the group members, to recognize the useful coping methods and strengths and to increase their use. In the fifth session; focuses on designing a positive future and steps towards achieving a positive future. In the sixth session, the sessions are summarized by the group leader and members.
  Interventions: Behavioral: Internet-Based Solution Focused Short-Term Group Counseling
- control group (Sham Comparator): A one-session nutrition education will be given to the control group. Students will be informed about the emotional eating behavior and they will be informed about the physical exercise and nutrition regulation process. Measurements will be repeated at the end of the session and 2 weeks later.
  Interventions: Other: healthy nutrition education

INTERVENTIONS:
Behavioral: Internet-Based Solution Focused Short-Term Group Counseling — Sessions will be held online once a week, with an average duration of 60-90 minutes, in the form of 6 sessions, via video-conference applications.
  Arms: experimental group
Other: healthy nutrition education — 60-minute single session healthy eating training
  Arms: control group

SUMMARY:
The study was carried out to determine the effect of internet-based solution-oriented group counseling on the emotional eating levels of nursing faculty students.

The population of the research of 481 nursing students studying at the Nursing Faculty in Istanbul. Sampling, on the other hand, is aimed at 60-person plans.

Within the scope of the study; At the 5% significance level and to be 16 in 1,204 domains, 32 individuals must be reached (df=30; t=1,697). Losses may occur before; Two experimental groups, each consisting of 15 students, and two control groups are targeted. The students will assigned to the experimental and control groups by simple random sampling method. The experimental group (n=26) will give solution-oriented group counseling on emotional eating once a week for 6 sessions over the internet. The control group (n=29) will trained 45-minute about healthy eating habits. Data will collected with the "Information Form", "Dutch Eating Behavior Questionnaire Emotional Eating Sub-Dimension" and "Challenges in Emotion Regulation Scale". The data will analies by chi-square test, independent groups t-test and repeated groups Anova test in SPSS program.

DETAILED DESCRIPTION:
Nutrition; It is the completion of the growth and development stages and the adequate intake of nutrients necessary for being healthy (Özmen et al. 2007). Maslow (1943) considers nutrition within the physiological needs at the first step in the hierarchy of needs and states that the purpose of satisfying physiological needs can also be the search for comfort and safety. Eating frequency and amount are also affected by emotions such as anxiety, anger, joy, depression, and sadness in addition to physiological hunger (Canetti et al. 2002). Emotional eating is expressed as a response to negative emotions and is seen as a way of regulating experienced negative emotions (Frayn & Knäuper, 2018). Bekker et al. (2004) reported that participants showed higher emotional eating behavior during negative affect compared to neutral mood periods. In addition, it is stated that impulsivity has an increasing effect on self-perceived emotional eating. In the study examining the effects of emotions on feeding behavior; anger has a higher effect on impulsive and emotional eating, and joy on hedonic eating compared to other emotions. It has also been reported that women tend to eat more emotionally during feelings of anger and sadness (Macht 1999). Studies indicate that individuals with high body mass index have more emotional eating behavior (Blair et al. 1990; Levoy et al. 2017). But Geliebter and Aversa. (2003) reported that emotional eating behavior is more common in normal-weight individuals in the face of positive emotions. In the study conducted with university students in the normal weight range; female students define stress, while male students define boredom and anxiety as factors that cause emotional eating behavior. It is observed that unhealthy foods are generally preferred during emotional eating and female students feel more guilty than males (Bennett et al. 2013). Considering that university students are in the transition stage to adulthood, healthy eating behaviors are of great importance (Mazıcıoğlu and Öztürk 2003). Nutritional behaviors of university students who are seen as a risky group in terms of nutritional problems (Pengpid and Peltzer 2018) and who are trying to adapt to a new order also affect their physical and mental health and academic performance (Ermiş et al. 2015). For the emotional eating behavior of university students, interventions focusing on emotion and stress management apart from dietary regulation are recommended (Bennett et al. 2013).

ELIGIBILITY:
Inclusion Criteria:

Having a higher score than the scale mean (DEBQ>20). To know Turkish.

Exclusion Criteria:

Having a mental or physical problem that prevents communication. Not attending more than two sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Internet-based solution-focused short-term group counseling has an effect on reducing the emotional eating levels of nursing students. | 2 months
  Çeviri sonuçları Solution-oriented group counseling applied online has a positive effect on the emotional eating levels of nursing students.
Internet-based solution-oriented short-term group counseling has an effect on reducing body mass indexes of nursing students. | 2 months
  Çeviri sonuçları Solution-oriented group counseling applied online has a positive effect on the emotional eating levels of nursing students.
Internet-based solution-oriented short-term group counseling has an effect on reducing the emotion regulation difficulties of nursing students. | 2 months
  Çeviri sonuçları Solution-oriented group counseling applied online has a positive effect on the emotional eating levels of nursing students.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Bekker MH, van de Meerendonk C, Mollerus J. Effects of negative mood induction and impulsivity on self-perceived emotional eating. Int J Eat Disord. 2004 Dec;36(4):461-9. doi: 10.1002/eat.20041. PMID 15558635
- [Background] Bennett J, Greene G, Schwartz-Barcott D. Perceptions of emotional eating behavior. A qualitative study of college students. Appetite. 2013 Jan;60(1):187-192. doi: 10.1016/j.appet.2012.09.023. Epub 2012 Oct 6. PMID 23046706
- [Background] Blair AJ, Lewis VJ, Booth DA. Does emotional eating interfere with success in attempts at weight control? Appetite. 1990 Oct;15(2):151-7. doi: 10.1016/0195-6663(90)90047-c. PMID 2268140
- [Background] Canetti L, Bachar E, Berry EM. Food and emotion. Behav Processes. 2002 Nov;60(2):157-164. doi: 10.1016/s0376-6357(02)00082-7. PMID 12426067
- [Background] Geliebter A, Aversa A. Emotional eating in overweight, normal weight, and underweight individuals. Eat Behav. 2003 Jan;3(4):341-7. doi: 10.1016/s1471-0153(02)00100-9. PMID 15000995
- [Background] Levoy E, Lazaridou A, Brewer J, Fulwiler C. An exploratory study of Mindfulness Based Stress Reduction for emotional eating. Appetite. 2017 Feb 1;109:124-130. doi: 10.1016/j.appet.2016.11.029. Epub 2016 Nov 24. PMID 27890474
- [Background] Pengpid S, Peltzer K. Risk of disordered eating attitudes and its relation to mental health among university students in ASEAN. Eat Weight Disord. 2018 Jun;23(3):349-355. doi: 10.1007/s40519-018-0507-0. Epub 2018 Apr 21. PMID 29681011